CLINICAL TRIAL: NCT06509893
Title: A Single-center, Randomized, 6-month, Non-inferiority Study to Compare the Safety and Efficacy of TICAgreLor mONotherapy Versus Dual Antiplatelet Therapy in Chronic Coronary Syndrome Patients Post Percutaneous Coronary IntErvention (TICALONE)
Brief Title: Ticagrelore Alone Post PCI
Acronym: TICALONE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Kojuri, professor, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IR.SUMS.MED.REC.1403.150
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous coronary intervention; dual antiplatelet therapy; clopidogrel; ticagrelor; MACE
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; Clopidogrel; Ticagrelor

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clopidogrel and aspirin (Active Comparator): Patients post PCI randomized to Aspirin 80 mg and clopidogrel 75 mg daily
  Interventions: Drug: aspirin 80 mg and clopidogrel 75 mg daily
- ticagrelor (Experimental): Patients post PCI randomized to Ticagrelor 90 mg PO two times daily
  Interventions: Drug: Ticagrelor 90 MG

INTERVENTIONS:
Drug: aspirin 80 mg and clopidogrel 75 mg daily — post PCI patients received these two drugs as dual antiplatelet regimen
  Arms: Clopidogrel and aspirin
Drug: Ticagrelor 90 MG — Post PCI patients receive Ticagrelor 90 mg two times daily as single potent antiplatelet
  Arms: ticagrelor

SUMMARY:
After PCI for CCS patients, single center double blind randomization will be done and patients will receive aspirin 80 mg and clopidogrel 75 mg versus 90 mg two times daily of ticagrelor, for 6 months and MACE will be followed in registry of professor Kojuri cardiology clinic

DETAILED DESCRIPTION:
An interventional cardiologist will perform angiography with the supervision of a fellow interventional cardiologist. Patients who need revascularization will undergo PCI using DES (Drug-eluting stent). PCI will be performed using the radial or femoral approach to achieve complete revascularization of at least one stenosis with a diameter of ≥50%. All target lesions will be revascularized using the 4th generation DES.

Randomization (1:1) will take place after diagnostic angiography but before stent insertion (figure 1). Eligible patients will be divided into two groups: the reference group, which will get conventional DAPT with aspirin and Clopidogrel (80 mg aspirin once daily, and 75mg clopidogrel once daily), and the experimental group, which will receive ticagrelor monotherapy (90mg twice daily) following PCI for six months.

Antiplatelet therapy will start before or at the time of PCI. Patients will receive a loading dose of assigned drugs (325mg for aspirin, 300mg for clopidogrel, and 180mg for ticagrelor) before stent insertion unless they are already on pre-PCI maintenance therapy with the mentioned drugs.

Subjects are randomly assigned a treatment strategy by an interactive web response system.

The primary efficacy endpoint is a composite of cardiac death, target vessel MI, stent thrombosis, and the need for revascularization occurring within 6 months of PCI. The secondary endpoints are all-cause death, occurrence of MACE including stroke (ischemic, hemorrhagic, or unknown), MI, arrhythmia, and each component of the primary endpoint at 6 months.

Safety is the third outcome

ELIGIBILITY:
Inclusion Criteria:

* Male or female above 20 years of age undergoing PCI with a drug-eluting stent for chronic coronary syndrome
* The patient has provided written informed consent as approved by the ethics committee of the Shiraz University of Medical Sciences.

Exclusion Criteria:

* Contraindication to aspirin, clopidogrel, ticagrelor, or any other reason that study drug should not be administered (including hypersensitivity, moderate or severe liver disease, active bleeding, and major surgery within 30 days)
* Atrial fibrillation or other indication for oral anticoagulant therapy.
* Concomitant oral or IV therapy with strong CYP3A inhibitors, CYP3A substrates with narrow therapeutic indices (cyclosporine, and quinidine), or strong CYP3A inducers ( rifampin, rifampicin, phenytoin, and carbamazepine)
* Females of child-bearing age unless negative pregnancy test at screening and willing to use effective contraception for the duration of trial
* Females who are breastfeeding at the time of enrolment.
* Unsuccessful PCI or PCI without optimal stent placement; this decision is made by the supervising interventional cardiologist.
* patients with anatomical SYNTAX score ≥23 prior to PCI
* Patients with planned surgical intervention to treat any cardiac or non-cardiac condition.
* Previous PCI in the last 6 months.
* Current (same hospitalization) or previous (within 12 months) acute coronary syndrome.
* History of definite stent thrombosis.
* Concomitant cardiac valve disease requiring invasive therapy.
* Acute heart failure.
* Active myocarditis.
* Cardiomyopathy.
* Patient in hemodialysis.
* History of stroke or transient ischemic cerebrovascular accident.
* History of intracranial hemorrhage or other intracranial pathology associated with increased bleeding risk.
* Hemoglobin <10 g/dL
* Peptic ulceration documented by endoscopy within the last 3 months unless healing proven by repeat endoscopy.
* Any other condition deemed by the investigator to place the patient at excessive risk of bleeding with ticagrelor.
* Participation in another trial with an investigational drug or device.
* Assessment that the subject is not likely to comply with the study procedures or have complete follow-up.
* Known drug or alcohol dependence within the past 12 months as judged by the investigator.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5400 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
stent thrombosis | 6 months
  Post PCI till 6 months any confirmed or suspected episodes of stent thrombosis based on ARCH definition
Major adverse cardiovascular events | 6 months
  Any episodes of myocardial infarction, acute coronary syndrome, revascularization, hospital admission and major vascular events will be recorded
Bleeding | 6 months
  any major or minor bleeding based on HASBLED criteria

SECONDARY OUTCOMES:
Treatment related adverse reactions | 6 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (2):
- Iran (2):
  - Cardiology Ward Shiraz University of Medical Sciences, Shiraz, Fars
  - professor Kojuroi cardiology clinic, Shiraz

IPD SHARING:
Plan to Share IPD: No
due to patients safety, data will be available on rational request

REFERENCES:
- [Derived] Mirhosseini SA, Akbari M, Aldavood D, Zarifkar H, Attar A, Kojuri J. Rationale and design of randomized non-inferiority clinical trial to compare the safety and efficacy of ticagrelor monotherapy with dual antiplatelet therapy in chronic coronary syndrome patients post percutaneous coronary intervention (TICALONE-TAHA10 Protocol). PLoS One. 2025 Jul 16;20(7):e0325663. doi: 10.1371/journal.pone.0325663. eCollection 2025. PMID 40668853